CLINICAL TRIAL: NCT06423976
Title: Collection of Clinical Material From Patients With Prostate Cancer or Undergoing Investigation for Diagnostic or Follow up Purposes for Molecular Characterisation and Microbiome Analysis
Brief Title: Microbiome Molecular Charaterisation
Acronym: MMC
Status: Recruiting | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5856
Record Dates: First submitted 2023-10-25; First posted 2024-05-21 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sequencing study — Sequencing of tumour samples for microbiome analysis and molecular charcterisation.

SUMMARY:
Preclinical models of prostate cancer have proved to be poorly predictive of the behaviour of the disease in patients. This protocol describes the acquisition of prostate cancer tissue or cells from patients with treatment naïve/hormone-sensitive and castration-resistant prostate cancer or patients undergoing diagnostic or follow up investigations. The knowledge gained will improve the investigators' understanding of the steps leading to the development of castration resistance and identify new molecular targets for treatment.

The human microbiome has been under investigation in a range of human diseases (i.e. metabolic disease/obesity, neurological disorders, cardiovascular disease, mental disorders, autoimmune disease, asthma and allergies) and cancer. The human microbiota can have direct (e.g. via direct genotoxicity, induction of chronic inflammation, etc.) and/or indirect (e.g. effects on tumour effects on tumour development or progression exerted through microbial communities that exist at a site distant to the tumour) effects on the disease. Emerging data supports the influence of the gut microbiota on the efficacy of anti-cancer treatments, including immunotherapy. To date, the impact of the gut microbiome on prostate cancer therapies is virtually unexplored. Based on the evidence to date, the investigators hypothesize that the gut flora may be altered by certain treatments for advanced prostate cancer, and that the composition of the microbiome in the gastrointestinal tract may be used to predict therapeutic efficacy or therapy-related toxicities; as well as prevent treatment toxicity and/or enhance treatment response.

Furthermore, the purpose is to investigate the association between gut flora and treatment response and related toxicities/morbidities in advanced prostate cancer.

DETAILED DESCRIPTION:
Prostate cancer is the second commonest malignancy in the UK and the second commonest cause of male mortality in the UK. Androgen deprivation therapy remains the mainstay of treatment, not only for advanced prostate cancer but also in the adjuvant and neo-adjuvant settings. Androgen deprivation therapy induces a remission in 80 to 90% of patients with advanced disease and results in a median progression-free survival of 12 to 33 months, at which time an androgen-independent phenotype usually emerges. This accounts for a median overall survival of 23 to 37 months from the initiation of androgen deprivation.

Recent preclinical studies have shown that the intestinal microbiota is associated with response to treatments such as platinum chemotherapy (oxaliplatin) [1], cyclophosphamide [2] and both CTLA-4 blockade [3] and anti-PD-L1 [4] immunotherapies. Eradication of commensal intestinal flora by antibiotic treatment, or via deriving specific-pathogen-free (SPF) and/or germ-free animals, has been shown to alter the therapeutic efficacy of these agents in tumour models. Intriguingly, a recent study in a melanoma model showed that responses to anti-PD-L1 immunotherapy could be increased by feeding animals a strain of Bifidobacterium - a species commonly used in probiotic supplements - prior to initiating therapy. Collectively, these studies suggest that the composition of the intestinal microbiome is both essential for therapeutic efficacy and a target that could potentially be modulated to enhance treatment response.

MMC is a prospective, observational, multi-centre study evaluating prostate cancer biology and associated microbiota.

Patients must be willing to undergo a fresh tumour biopsy for molecular analyses. Following consent to MMC, fresh tumour tissue will be sent to designated research laboratories (see laboratory manual) for analyses to identify molecular aberrations and dysbiosis through targeted or broader molecular analyses (e.g. exome, transcriptome, whole genome), as well as (when indicated) orthogonal assays (e.g. immunohistochemistry, immunofluorescence, RNAish, digital droplet PCR). MMC will focus on tumour and microbiota characterisation (both CSPC and mCRPC) with recent studies indicating that this is a highly heterogeneous disease. The data acquired will be made available to patients, when indicated, and their clinical care team to help select what early clinical trial options merit consideration.

Patients will not receive any treatment or IMP as part of this MMC protocol. Results of the molecular characterisation and microbiota studies will be made available to the treating investigator and the patient at a study specific visit (telephonic or face-to-face); patients will then be followed up every 6-months via medical notes review or telephone for survival and anti-cancer treatment data.

ELIGIBILITY:
Inclusion Criteria:

1. Male >=18 years.
2. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 - 2.
3. Undergoing investigation for diagnosis, or with a proven diagnosis of prostate cancer and undergoing further investigation or clinical trial participation.
4. Patients with tumour deemed by the designated investigator as safely suitable for fresh biopsy AND who are medically fit (according to local practice) to undergo a biopsy or surgical procedure to acquire tumour tissue.
5. Willing and able to comply with the requirements of the sample collection including fresh tumour biopsy.
6. The subject is capable of understanding and complying with the protocol requirements and has given written informed consent.
7. A record of PSA levels within last 3 months.

Exclusion Criteria:

1. The presence of any haematological disorders, including coagulation disorders, which would be a contraindication if patient were to undergo a biopsy.
2. Any psychiatric illness/social situations that would limit compliance with study requirements.
3. Presence of any concurrent condition or situation, which, in the investigator's opinion, may put the patient at significant risk, may confound the study results, or may interfere significantly with the patient's participation in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample size is not based on formal statistical power analyses but rather on pragmatic and feasibility considerations. Our experience with our previous MC study lets us assume that we will be able to recruit 200 patients per year (from 1-2 participating centres) over a recruitment period of five years. Thus, the total expected sample size will be 1000 patients. The expected study endpoint analysis will commence following the 5-year recruitment period but no longer than the overall 15-year end of study timeline.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2038-10 (Estimated); Study Completion 2038-10 (Estimated)

PRIMARY OUTCOMES:
Microbiome composition in prostate cancer patients | through study completion, an average of 1 year
  Describing the microbiome composition in prostate cancer patients using metagenomic and metabolomic studies.

SECONDARY OUTCOMES:
Prevalence of prostate cancer aberrations | through study completion, an average of 1 year
  Prevalence of prostate cancer aberrations including at DNA, RNA, protein or metabolite level.
Patient clinical outcomes | time to castration resistance, time to treatment progression and overall survival.
  Overall response rate defined as the proportion of patients with partial or complete response to a given treatment according to clinical [Symptoms], biochemical [PSA] or radiographic criteria (e.g., RECIST).
  * Prognostic clinical parameters - Hb [Haemoglobin], Albumin, LDH & ALP
  * Time to castration resistance defined as time from study entry to diagnosis of castration resistant prostate cancer.
  * Time to treatment progression defined as time from start of therapy to progression (clinical [Symptoms], biochemical [PSA], or radiographic) on treatment.
  * Progression-free survival defined as the time from start of treatment to progression on treatment (clinical [Symptoms], biochemical [PSA] or radiographic) or death from any cause.
  * Overall survival defined as time from study entry to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Johann De-Bono, Principal Investigator — The Royal Marsden NHS FT\The Institute of Cancer Research
Locations (1):
- Institute of Cancer Research/Royal Marsden NHS FT, Sutton, Surrey, United Kingdom